CLINICAL TRIAL: NCT03312881
Title: Characterisation of Neuropathic Pain in Children: Multimodal Assessment and Diagnosis
Brief Title: Neuropathic Pain in Children: Multimodal Assessment and Diagnosis
Status: Completed | Type: Observational
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Other Study IDs: 17NC03
Record Dates: First submitted 2017-09-27; First posted 2017-10-18 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Neuropathic Pain; Child, Only
Keywords: pain; neuropathic; children; QST
MeSH Terms: conditions — Neuralgia; Pain | interventions — Neuroimaging; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neuropathic pain: Children with clinical diagnosis of neuropathic pain. Interventions: patient reported outcome measures, quantitative sensory testing, neuroimaging
  Interventions: Diagnostic Test: quantitative sensory testing; Diagnostic Test: neuroimaging; Other: Patient Reported Outcome Measures
- non-neuropathic pain: Children with clinical diagnosis of non-neuropathic pain. Interventions: patient reported outcome measures
  Interventions: Other: Patient Reported Outcome Measures

INTERVENTIONS:
Diagnostic Test: quantitative sensory testing — multiple modality testing of generalized and localized changes in somatosensory perception
  Groups: neuropathic pain
Diagnostic Test: neuroimaging — magnetic resonance imaging (MRI)
  Groups: neuropathic pain
Other: Patient Reported Outcome Measures — neuropathic pain screening tool; validated questionnaires

SUMMARY:
Some children experience chronic pain that is related to damage or diseases that affect the nerves that send pain signals. This is known as neuropathic pain. This is not well understood and can be difficult to diagnose. It can often produce unusual feelings such as sensitivity of the skin to light touch. Neuropathic pain is often severe and difficult to treat, and can affect quality of life for the child and family. This study aims to better characterise the symptoms and signs, and impact of neuropathic pain in children.

DETAILED DESCRIPTION:
The Investigators will determine whether a questionnaire to identify neuropathic pain in adults is also useful in children. This will help paediatricians and other doctors to recognise neuropathic pain and start appropriate treatment or know when to refer children to a chronic pain clinic.The Investigators will also measure the effects of neuropathic pain on mood, sleep, and quality of life (using questionnaires); identify changes in the sensitivity of the skin to touch and other sensations (using specialised sensory tests); and determine the feasibility of brain imaging for assessing changes in the brain (using magnetic resonance imaging or MRI), in children with neuropathic pain. This information will allow the investigators to measure how effective different types of treatment are, and help ensure children get the most appropriate treatment or interventions to reduce pain and effects on quality of life.

This pilot study of 10-18 year olds diagnosed with neuropathic pain will involve completion of questionnaires by the child and parent, and sensory testing in the child, after their clinic appointment. For some families, there will be an additional visit for MRI. Children will be recruited from the Chronic Pain Outpatients service at Great Ormond Street Hospital NHS Trust. This research is funded by Great Ormond Street Hospital Children's Charity.

ELIGIBILITY:
Inclusion Criteria:

* children with a clinical diagnosis of chronic neuropathic pain for the full protocol
* children with a clinical diagnosis of non-neuropathic origin for S-LANSS validation and questionnaires
* children aged 10-18 years

Exclusion Criteria:

* significant impairment of comprehension (less than school level for 10 year old) that will limit understanding of sensory testing instructions
* inadequate english language skills as questionnaires are validated in English and sensory testing instructions can only be delivered by the Investigators in English For brain imaging, patients will be excluded if they have
* significant medical illness or other (non-neuropathic) neurological disease
* pregnancy
* magnetic implants of any type.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will recruit children and adolescents aged 10-18 years referred to the Great Ormond Street Hospital Pain Service who are clinically diagnosed as having neuropathic pain.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Self-Report Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) questionnaire | 3 years
  Sensitivity and specificity of a neuropathic screening tool in children; includes 5 questions related to symptoms and pain descriptors and 2 related to examination

SECONDARY OUTCOMES:
Paediatric Quality of Life Inventory (Child and Parent report) | 3 years
  evaluates 23 items relating to the child's functioning in four dimensions: physical; emotional; social; and school.
Pain Catastrophizing Scale (Child and Parent versions) | 3 years
  13 items assessing 3 aspects of pain experience: the tendency to magnify the threat value of pain (magnification), to feel helpless in the context of pain (helplessness), and to worry about it more (rumination)
Pain Coping Questionnaire | 3 years
  comprises 39 items relating to information seeking; problem solving; seeking social support; positive self-statements; behavioural distraction; cognitive distraction; externalising; and internalising/catastrophizing
Adolescent Sleep-Wake Scale-Revised | 3 years
  evaluates 10 items relating to: falling asleep and reinitiating sleep; returning to wakefulness; and going to bed
Paediatric Index of Emotional Distress | 3 years
  comprises 14 items related to symptoms of anxiety and depression, with a maximum score of 42
Hospital Anxiety and Depression Scale | 3 years
  measures anxiety and depression in adults (parents) and comprises 14 items
Quantitative Sensory Testing | 3 years
  Sensory profile in terms of gain or loss of sensitivity
Magnetic Resonance Imaging | 3 years
  pilot study to assess feasibility and acceptability of MRI in this patient group

CONTACTS AND LOCATIONS:
Overall Officials: Suellen M Wallker, MBBS PhD, Principal Investigator — UCL GOS Institute of Child Health
Locations (1):
- IChildHealth, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Walker SM, Peters J, Verriotis M, Farag F, Jay MA, Howard RF. Sensitivity and Specificity of a Neuropathic Screening Tool (Self-Report Leeds Assessment of Neuropathic Symptoms and Signs, S-LANSS) in Adolescents With Moderate-Severe Chronic Pain. J Pain. 2024 Feb;25(2):451-465. doi: 10.1016/j.jpain.2023.09.006. Epub 2023 Sep 21. PMID 37741521
- [Derived] Verriotis M, Peters J, Sorger C, Walker SM. Phenotyping peripheral neuropathic pain in male and female adolescents: pain descriptors, somatosensory profiles, conditioned pain modulation, and child-parent reported disability. Pain. 2021 Jun 1;162(6):1732-1748. doi: 10.1097/j.pain.0000000000002172. PMID 33394878

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT03312881/Prot_SAP_000.pdf